CLINICAL TRIAL: NCT05893797
Title: Assessment of Participant Adherence and Glucose Control While Using a Connected Insulin Management Platform
Brief Title: A Study of LY8888AX in Participants Using a Connected Insulin Management Platform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18171; F3Z-MC-IORW (Other: Eli Lilly and Company); 2022-A02807-36 (Other: EU Trial Number)
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes; Type 2 Diabetes Treated With Insulin
Keywords: T1D; T2D
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Humalog Tempo Pen With CGM Monitoring (Experimental): Study Period 1: Weeks 1 to 6
  * Participants used a Sponsor-provided Humalog Tempo Pen with Tempo Smart Button (TSB), Dexcom G6 continuous glucose monitoring (CGM), and the Glooko Research Mobile App (RMA) to share insulin dose and timing data with healthcare providers (HCPs) via the Glooko HCP platform. Mealtime insulin data was masked to participants but visible to HCPs. Participants followed their usual insulin regimen and lifestyle, manually logged basal insulin and activities in the app. After 6 weeks, data was unmasked and reviewed with HCPs.
  Study Period 2: Weeks 7 to 18
  * Participants used the Humalog Tempo Pen with TSB, Dexcom G6 CGM, and Glooko RMA study app for 12 weeks. Insulin dose and timing data was unmasked and visible to both participants and HCPs via the Glooko RMA and HCP platform. Participants regularly upload CGM and pen data. HCPs monitor adherence and follow up as needed to ensure data transfer and CGM use.
  Interventions: Drug: Insulin Lispro; Device: Tempo Smart Button; Device: Dexcom G6 CGM; Device: Glooko Research Mobile App (RMA)

INTERVENTIONS:
Drug: Insulin Lispro — As prescribed.
  Other Names: Humalog Tempo Pen
Device: Tempo Smart Button — Attached to the Tempo Pen
Device: Dexcom G6 CGM — Continuous glucose monitor
Device: Glooko Research Mobile App (RMA) — Installed on a study provided android phone.

SUMMARY:
The main purpose of this study is to assess participant adherence and glucose control while using a connected insulin management platform. Approximately 50 participants will be enrolled in each country.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed (clinically) with T1D for at least 1 year or are patients with T2D on basal bolus insulin therapy for at least 6 months
* HbA1c ≥8% as confirmed by point-of-care test at screening
* Are currently using the Dexcom G6 CGM or agree to start using the Dexcom G6 during the study and agree to switch to Glooko RMA
* Are currently using Humalog ® insulin or another rapid acting insulin analogue (e.g., Apidra® , or Novorapid ® ) and agree to switch to study-provided Humalog mealtime insulin for duration of trial
* Have been prescribed ≥3 doses of bolus insulin per day
* Must be taking a stable insulin dose regimen (per investigator's judgement) for at least 3 months preceding study screening
* Have in-home refrigeration for storage of insulin

Exclusion Criteria:

* Previously used the Glooko RMA and/or Dexcom G6 CGM and were judged by the investigator to be non-adherent
* Have participated, within the last 30 days, in a clinical study involving an investigational product. If the previous investigational product has a long half-life, 5 half-lives or 30 days (whichever is longer) should have passed
* Have previously used or have been using an approved or investigational connected pen system within the 3 months prior to screening
* Are currently breastfeeding, pregnant, or plan to become pregnant during the next 4-6 months
* Are on ultra-rapid insulin (e.g., Fiasp or Lyumjev) or rapid acting human insulin (i.e., Humulin) for previous 3 months, at the time of screening
* Are currently undergoing dialysis treatment or have any other medical condition which may preclude them from participating in this trial as per the investigator's judgement
* Have vision loss or vision impairment that does not allow recognition of Glooko RMA screen features

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (9):
- France (9):
  - CHU Strasbourg-Hautepierre, Strasbourg, Alsace
  - CHU de Caen Hôpital Cote de Nacre, Caen, Cedex 9
  - CHU de Besancon Hopital Jean Minjoz, Besançon
  - Centre Hospitalier Sud Francilien-Pharmacie, Corbeil-Essonnes
  - Chu de Grenoble, Grenoble Cédex 9
  - CHU de Lyon, Lyon
  - CHU - l'Assistance Publique - Hôpitaux de Marseille, Marseille
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet, Nice
  - Groupe Hospitalier Mutualiste Les Portes du Sud, Vénissieux

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 36 participants were enrolled in the study, defined as those who provided informed consent and met eligibility criteria. Additionally, 49 healthcare providers (HCPs) consisting of principal investigator, study coordinator or nurse associated with this study were only surveyed regarding certain study outcomes specific to HCP questionnaires. As per prespecified study design HCPs were not enrolled in the study.
Pre-assignment Details: Of the 49 HCPs, 37 completed at least one post-baseline questionnaire assessing device preference, satisfaction, and usefulness. HCP responses were collected as part of a pre-specified endpoint and data represent independent evaluations, are not linked to any specific participant.
Period: Study Period 1 (Weeks 1 to 6)
Arm/Group | Humalog Tempo Pen With CGM Monitoring
Started | 36
Main Analysis Set (Main Analysis set: * Participants with at least 10 valid CGM days out of the last 14 days in the study period 1 (masked) in Week 5 and week 6.) | 25
Number of HCPs Surveyed for Study Outcomes Specific to HCP Questionnaires | 49
Completed | 32
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2
Period: Study Period 2 (Weeks 7 to 18)
Arm/Group | Humalog Tempo Pen With CGM Monitoring
Started | 32
Main Analysis Set (Main Analysis set: * Participants with at least 20 of 28 valid CGM days during study period 2 in weeks 15 to 18 or if discontinued early that have at least 20 valid CGM days in the whole study period 2/week 7 to 18.) | 24
Completed | 30
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Arm/Group | Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  France | 36
Type of diabetes diagnosed [Count of Participants; unit: Participants]
  Type 1 diabetes mellitus | 20
  Type 2 diabetes mellitus | 16
Diabetes duration [Mean (Standard Deviation); unit: years] | 20.06 (9.12)

OUTCOME MEASURES:

1. Primary Outcome: Number of Missed Bolus Doses (MBDs) Per Week
Description: Missed bolus dose is defined as no insulin dose from 1 hour prior to through 1 hour after the start of a glucose excursion (meal), where a glucose excursion was defined as a greater than (>) 70 milligrams per deciliter (mg/dL) (>3.9 millimoles per liter [mmol/L]) rise within 2 hours, not preceded by a value <70 mg/dL (<3.9 mmol/L).
Time Frame: Study Period 1: Week 6 ; Study Period 2: Week 18
Population: All participants from main analysis set who had evaluable data for this outcome.
Measure: Mean (Standard Deviation); unit: missed bolus dose per week
Groups:
- Study Period 1 - Humalog Tempo Pen With CGM Monitoring: Study Period 1: Weeks 1 to 6
  * Participants used a Sponsor-provided Humalog Tempo Pen with Tempo Smart Button (TSB), Dexcom G6 continuous glucose monitoring (CGM), and the Glooko Research Mobile App (RMA) to share insulin dose and timing data with healthcare providers (HCPs) via the Glooko HCP platform. Mealtime insulin data was masked to participants but visible to HCPs. Participants followed their usual insulin regimen and lifestyle, manually logged basal insulin and activities in the app. After 6 weeks, data was unmasked and reviewed with HCPs.
- Study Period 2 - Humalog Tempo Pen With CGM Monitoring: Study Period 2: Weeks 7 to 18
  * Participants used the Humalog Tempo Pen with TSB, Dexcom G6 CGM, and Glooko RMA study app for 12 weeks. Insulin dose and timing data was unmasked and visible to both participants and HCPs via the Glooko RMA and HCP platform. Participants regularly upload CGM and pen data. HCPs monitor adherence and follow up as needed to ensure data transfer and CGM use.
Arm/Group | Study Period 1 - Humalog Tempo Pen With CGM Monitoring | Study Period 2 - Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 25 | 24
missed bolus dose per week | 2.3 (2.29) | 2.3 (1.56)

2. Secondary Outcome: Percentage of Time in Blood Glucose (BG) Range 70 to 180 mg/dL Captured by Continuous Glucose Monitoring (CGM)
Time Frame: Study Period 1: Week 6; Study Period 2: Week 18
Population: All participants from main analysis set who had evaluable data for this outcome.
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | Study Period 1 - Humalog Tempo Pen With CGM Monitoring | Study Period 2 - Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 25 | 24
Percentage of Time | 43.1 (17.17) | 41.6 (17.76)

3. Secondary Outcome: Percentage of Time in Hyperglycemic Range of >180 mg/dL and >250 mg/dL Captured by CGM
Time Frame: Study Period 1: Week 6; Study Period 2: Week 18
Population: All participants from main analysis set who had evaluable data for this outcome.
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | Study Period 1 - Humalog Tempo Pen With CGM Monitoring | Study Period 2 - Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 25 | 24
Percentage of Time
  >180 mg/dL | 56 (17.22) | 57.5 (17.89)
  >250 mg/dL | 24.7 (17.91) | 26.3 (17.76)

4. Secondary Outcome: Percentage of Time in Hypoglycemic Range <54 mg/dL and 54 to 69 mg/dL Captured by CGM
Time Frame: Study Period 1: Week 6; Study Period 2: Week 18
Population: All participants from main analysis set who had evaluable data for this outcome.
Measure: Mean (Standard Deviation); unit: Percentage of Time
Arm/Group | Study Period 1 - Humalog Tempo Pen With CGM Monitoring | Study Period 2 - Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 25 | 24
Percentage of Time
  <54 mg/dL | 0.2 (0.39) | 0.2 (0.43)
  54 to 69 mg/dL | 0.7 (0.67) | 0.7 (0.79)

5. Secondary Outcome: Coefficient of Variation for Glucose
Time Frame: Study Period 1: Week 6; Study Period 2: Week 18
Population: All participants from main analysis set who had evaluable data for this outcome.
Measure: Mean (Standard Deviation); unit: percentage of coefficient of variation
Arm/Group | Study Period 1 - Humalog Tempo Pen With CGM Monitoring | Study Period 2 - Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 25 | 24
percentage of coefficient of variation | 28.8 (5.82) | 28.9 (6.13)

6. Secondary Outcome: Mean Glucose as Measured by CGM
Time Frame: Study Period 1: Week 6; Study Period 2: Week 18
Population: All participants from main analysis set who had evaluable data for this outcome.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Study Period 1 - Humalog Tempo Pen With CGM Monitoring | Study Period 2 - Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 25 | 24
mg/dL | 202.8 (33.18) | 206 (35.44)

7. Secondary Outcome: Number of Mistimed Bolus Dose Per Week
Description: A mistimed bolus dose is defined as a bolus dose administered from the start of a glucose excursion up to 1 hour after the start of glucose excursion and before the peak of glucose excursion.
Time Frame: Study Period 1: Week 6 ; Study Period 2: Week 18
Population: All participants from main analysis set who had evaluable data for this outcome.
Measure: Mean (Standard Deviation); unit: Mistimed bolus dose per week
Arm/Group | Study Period 1 - Humalog Tempo Pen With CGM Monitoring | Study Period 2 - Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 25 | 24
Mistimed bolus dose per week | 3.1 (2.02) | 2.6 (1.55)

8. Secondary Outcome: Total Insulin Dose Per Day
Time Frame: Study Period 1: Week 6; Study Period 2: Weeks 18
Population: All participants from main analysis set who had evaluable data for this outcome.
Measure: Mean (Standard Deviation); unit: Total insulin units per day
Arm/Group | Study Period 1 - Humalog Tempo Pen With CGM Monitoring | Study Period 2 - Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 25 | 24
Total insulin units per day | 61.6 (57.75) | 60.8 (51.56)

9. Secondary Outcome: Number of Correction Bolus Dose Per Week
Description: Correction bolus is defined as taking a bolus dose given after the peak of a glucose excursion but within 4 hours from the start of a glucose excursion and prior to start of next glucose excursion.
Time Frame: Study Period 1: Week 6; Study Period 2: Week 18
Population: All participants from main analysis set who had evaluable data for this outcome.
Measure: Mean (Standard Deviation); unit: Correction bolus dose per week
Arm/Group | Study Period 1 - Humalog Tempo Pen With CGM Monitoring | Study Period 2 - Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 25 | 24
Correction bolus dose per week | 2.4 (1.73) | 2.6 (1.6)

10. Secondary Outcome: Correlation Between Missed Bolus Dose and Glycemic Outcomes [i.e., HbA1c, Time in BG Range (70-180 mg/dL), Time in Hyperglycemic Range (>250 mg/dL), and Time in Hypoglycemia (<54 mg/dL)] Using Raw CGM Integrated Data From Tempo Pen and Tempo Smart Button
Description: Correlation between Missed Bolus Dose and Glycemic Outcomes i.e., HbA1c, Time in Blood glucose (BG) Range (70-180 mg/dL), Time in Hyperglycemic Range (>250 mg/dL), and Time in Hypoglycemia (<54 mg/dL) was calculated by spearman correlation. Spearman correlation coefficients range from -1 to +1. A value of -1 indicates a perfect negative correlation, and +1 indicates a perfect positive correlation.
Time Frame: Study Period 1: Week 6; Study Period 2: Week 18
Population: All participants from main analysis set who had evaluable data for this outcome. Number analyzed are the participants who were evaluable for the given categories.
Measure: Number; unit: Correlation coefficient
Arm/Group | Study Period 1 - Humalog Tempo Pen With CGM Monitoring | Study Period 2 - Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 25 | 24
Correlation coefficient
  HbA1c: number analyzed (Participants) | 25 | 23
  HbA1c | -0.084 | -0.058
  Time in BG Range (70-180 mg/dL) | 0.175 | -0.111
  Time in Hyperglycemic Range (>250 mg/dL) | -0.217 | 0.156
  Time in Hypoglycemia Range (<54 mg/dL) | 0.068 | 0.079

11. Secondary Outcome: Correlation Between Mistimed Bolus Dose and Glycemic Outcomes [i.e., HbA1c, Time in BG Range (70-180 mg/dL), Time in Hyperglycemic Range (>250 mg/dL), Time in Hypoglycemia (<54 mg/dL)] Using Raw CGM Integrated Data From Tempo Pen and Tempo Smart Button
Description: Correlation between Mistimed Bolus Dose and Glycemic Outcomes i.e., HbA1c, Time in Blood glucose (BG) Range (70-180 mg/dL), Time in Hyperglycemic Range (>250 mg/dL), and Time in Hypoglycemia (<54 mg/dL) was calculated by spearman correlation. Spearman correlation coefficients range from -1 to +1. A value of -1 indicates a perfect negative correlation, and +1 indicates a perfect positive correlation.
Time Frame: Study Period 1: Week 6; Study Period 2: Week 18
Population: as for outcome 10
Measure: Number; unit: Correlation coefficient
Arm/Group | Study Period 1 - Humalog Tempo Pen With CGM Monitoring | Study Period 2 - Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 25 | 24
Correlation coefficient
  HBa1C: number analyzed (Participants) | 25 | 23
  HBa1C | -0.132 | -0.150
  Time in BG Range (70-180 mg/dL) | 0.139 | 0.020
  Time in Hyperglycemic Range (>250 mg/dL) | -0.082 | -0.054
  Time in Hypoglycemia (<54 mg/dL) | -0.203 | -0.060

12. Secondary Outcome: Study Period 1: Participant Questionnaires (Device Satisfaction)- On Average, How Satisfied Are You With Your Current Insulin Pen?
Description: Participant questionnaires evaluated responses to the Humalog Tempo Pen and Tempo smart button device focusing on platform satisfaction, preferences, and usefulness.
  To assess existing device satisfaction of tempo pen and smart button that participants were using before the study, participants were asked: "On average, how satisfied are you with your current insulin pen?" Participants were categorized based on their responses on a 5-point Likert scale as below and are reported
  1. Extremely Unsatisfied
  2. Unsatisfied
  3. Neutral
  4. Satisfied
  5. Extremely Satisfied
Time Frame: At Baseline
Population: Study period 1: All participants from main analysis set who had evaluable data for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Period 1 - Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 25
Participants
  Extremely unsatisfied | 0
  Unsatisfied | 1
  Neutral | 5
  Satisfied | 10
  Extremely satisfied | 9

13. Secondary Outcome: Study Period 1: Participant Questionnaires (Device Satisfaction) - On Average, How Satisfied Are You With the Way You Manage Your Insulin Treatment on a Day-to-day Basis?
Description: Participant questionnaires evaluated responses to the Humalog Tempo Pen and Tempo smart button device focusing on platform satisfaction, preferences, and usefulness.
  To assess existing device satisfaction of tempo pen and smart button that participants were using before the study, participants were asked: "On average, how satisfied are you with the way you manage your insulin treatment on a day-to-day basis?" Participants were categorized based on their responses on a 5-point Likert scale as below and are reported.
  1. Extremely Unsatisfied
  2. Unsatisfied
  3. Neutral
  4. Satisfied
  5. Extremely Satisfied
Time Frame: At Baseline
Population: Study period 1: All participants from main analysis set who had evaluable data for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Period 1 - Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 25
Participants
  Extremely unsatisfied | 3
  Unsatisfied | 2
  Neutral | 9
  Satisfied | 8
  Extremely satisfied | 3

14. Secondary Outcome: Study Period 2: Participant Questionnaires (Device Preference) - I Prefer the Connected Insulin Pen Compared to the Insulin Pen I Used Before the Study?
Description: Participant questionnaires evaluated responses to the Humalog Tempo Pen and Tempo smart button device focusing on platform satisfaction, preferences, and usefulness.
  To assess device preference of Humalog Tempo Pen and Tempo smart button participants were asked: "I prefer the connected insulin pen compared to the insulin pen I used before the study?" Participants were categorized based on their responses on a 5-point Likert scale as below and are reported
  1. Strongly disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly agree
Time Frame: Study Period 2: Week 18
Population: Study period 2: All participants from main analysis set who had evaluable data for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Period 2 - Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 25
Participants
  Strongly disagree | 1
  Disagree | 3
  Neutral | 4
  Agree | 8
  Strongly agree | 9

15. Secondary Outcome: Study Period 2: Participant Questionnaires (Device Usefulness) - I Found the App Difficult to Use to Monitor my Insulin Doses
Description: Participant questionnaires evaluated responses to the Humalog Tempo Pen and Tempo smart button device focusing on satisfaction, preferences, and usefulness.
  To assess device usefulness of Humalog Tempo Pen and Tempo smart button participants were asked: "I found the app difficult to use to monitor my insulin doses" Participants were categorized based on their responses on a 5-point Likert scale as below and are reported.
  1. Strongly Disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree
Time Frame: Study Period 2: Week 18
Population: Study period 2: All participants from main analysis set who had evaluable data for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Period 2 - Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 25
Participants
  Strongly Disagree | 9
  Disagree | 10
  Neutral | 3
  Agree | 3
  Strongly Agree | 0

16. Secondary Outcome: Study Period 2: Participant Questionnaires (Device Usefulness) - It Helped me to Forget Fewer Doses
Description: Participant questionnaires evaluated responses to the Humalog Tempo Pen and Tempo smart button device focusing on platform satisfaction, preferences, and usefulness.
  To assess device usefulness of Humalog Tempo Pen and Tempo smart button participants were asked: "It helped me to forget fewer doses" Participants were categorized based on their responses on a 5-point Likert scale as below and are reported
  1. Strongly Disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree
Time Frame: Study Period 2: Week 18
Population: Study period 2: All participants from main analysis set who had evaluable data for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Period 2 - Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 25
Participants
  Strongly Disagree | 5
  Disagree | 1
  Neutral | 7
  Agree | 6
  Strongly Agree | 6

17. Secondary Outcome: Study Period 2: Participant Questionnaires (Device Usefulness) - I no Longer Had to Worry About When my Last Dose Was Injected or Not
Description: Participant questionnaires evaluated responses to the Humalog Tempo Pen and Tempo smart button device focusing on platform satisfaction, preferences, and usefulness.
  To assess device usefulness of Humalog Tempo Pen and Tempo smart button participants were asked "I no longer had to worry about when my last dose was injected or not" Participants were categorized based on their responses on a 5-point Likert scale as below and are reported
  1. Strongly Disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree
Time Frame: Study Period 2: Week 18
Population: Study period 2: All participants from main analysis set who had evaluable data for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Period 2 - Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 25
Participants
  Strongly Disagree | 3
  Disagree | 4
  Neutral | 2
  Agree | 7
  Strongly Agree | 9

18. Secondary Outcome: Study Period 2: Participant Questionnaires (Device Usefulness) - Having All my Insulin and Glucose Data in One Place Simplified my Diabetes Management
Description: Participant questionnaires evaluated responses to the Humalog Tempo Pen and Tempo smart button device focusing on platform satisfaction, preferences, and usefulness.
  To assess device usefulness of Humalog Tempo Pen and Tempo smart button participants were asked: "Having all my insulin and glucose data in one place simplified my diabetes management" Participants were categorized based on their responses on a 5-point Likert scale as below and are reported
  1. Strongly Disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree
Time Frame: Study Period 2: Week 18
Population: Study period 2: All participants from main analysis set who had evaluable data for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Period 2 - Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 25
Participants
  Strongly Disagree | 1
  Disagree | 1
  Neutral | 6
  Agree | 9
  Strongly Agree | 8

19. Secondary Outcome: Study Period 2: Participant Questionnaires (Device Usefulness): I Found the Connected Pen to be Difficult to Use
Description: Participant questionnaires evaluated responses to the Humalog Tempo Pen and Tempo smart button device focusing on platform satisfaction, preferences, and usefulness.
  To assess device usefulness of Humalog Tempo Pen and Tempo smart button participants were asked: "I found the connected pen to be difficult to use" Participants were categorized based on their responses on a 5-point Likert scale as below and are reported.
  1. Strongly Disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree
Time Frame: Study Period 2: Week 18
Population: Study period 2: All participants from main analysis set who had evaluable data for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Period 2 - Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 25
Participants
  Strongly Disagree | 13
  Disagree | 7
  Neutral | 3
  Agree | 2
  Strongly Agree | 0

20. Secondary Outcome: Study Period 2: Participant Questionnaires (Device Usefulness): The Use of the Connected Insulin Pen Reduced the Amount of Time I Spent on my Diabetes Management
Description: Participant questionnaires evaluated responses to the Humalog Tempo Pen and Tempo smart button device focusing on platform satisfaction, preferences, and usefulness.
  To assess device usefulness of Humalog Tempo Pen and Tempo smart button participants were asked: "The use of the connected insulin pen reduced the amount of time I spent on my diabetes management". Participants were categorized based on their responses on a 5-point Likert scale as below and are reported.
  1. Strongly Disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree
Time Frame: Study Period 2: Week 18
Population: Study period 2: All participants from main analysis set who had evaluable data for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Period 2 - Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 25
Participants
  Strongly Disagree | 6
  Disagree | 5
  Neutral | 5
  Agree | 5
  Strongly Agree | 4

21. Secondary Outcome: Health Care Provider (HCP) Questionnaires (Device Satisfaction) - On Average, How Satisfied Are You With the Connected Insulin Pen Your Patients Have Been Using in the Study?
Description: The Health Care Provider (HCP) questionnaires evaluated responses from HCPs related to Humalog Tempo Pen and Tempo smart button device focusing on satisfaction, preferences, and usefulness. Questionnaire was completed independently by HCPs (Including Principal Investigator, study coordinator or nurse). This evaluation was a general, aggregate assessment and was not linked to any specific participant. To assess Humalog Tempo Pen and Tempo smart button device satisfaction HCPs were asked: "On average, how satisfied are you with the connected insulin pen your patients have been using in the study?"
  HCPs were categorized based on their responses on a 5-point Likert scale as below and are reported.
  1. Extremely Unsatisfied
  2. Unsatisfied
  3. Neutral
  4. Satisfied
  5. Extremely Satisfied
Time Frame: Following completion of participant's Last visit in the study (approximately 3 days after last visit on week 18)
Population: All Health Care Providers (HCPs) who completed at least one question on the post baseline HCP questionnaire following completion of participant's last visit in the study. Overall Number of Participants Analyzed are the HCPs who provided responses to the HCP questionnaire and not the study participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 37
Participants
  Extremely Unsatisfied | 3
  Unsatisfied | 11
  Neutral | 14
  Satisfied | 7
  Extremely satisfied | 2

22. Secondary Outcome: Health Care Provider (HCP) Questionnaires (Device Usefulness) - Offered me Objective Date on my Patients Dosing History Allowing me to Provide Appropriate Dosing Guidance
Description: The Health Care Provider (HCP) questionnaires evaluated responses from HCPs related to Humalog Tempo Pen and Tempo smart button device focusing on device satisfaction, preferences, and usefulness. Questionnaire was completed independently by HCPs (including principal Investigator, study coordinator or nurse). This evaluation was a general, aggregate assessment and was not linked to any specific participant. To assess Humalog Tempo Pen and Tempo smart button device usefulness HCPs were asked: "Offered me objective date on my patients dosing history allowing me to provide appropriate dosing guidance".
  HCPs were categorized based on their responses on a 5-point Likert scale as below and are reported.
  1. Strongly Disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree
Time Frame: Following completion of participant's Last visit in the study (approximately 3 days after last visit on week 18)
Population: All Health Care Providers (HCPs) who completed at least one question on the post-baseline HCP questionnaire following completion of participant's last visit in the study. Overall Number of Participants Analyzed are the HCPs who provided responses to the HCP questionnaire and not the study participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 37
Participants
  Strongly Disagree | 1
  Disagree | 3
  Neutral | 10
  Agree | 18
  Strongly Agree | 5

23. Secondary Outcome: Health Care Provider (HCP) Questionnaires (Device Usefulness)- It Improved my Confidence in Making Appropriate Dosing Decisions
Description: The Health Care Provider (HCP) questionnaires evaluated responses from HCPs related to Humalog Tempo Pen and Tempo smart button device focusing on satisfaction, preferences, and usefulness.
  Questionnaire was completed independently by HCPs (including principal Investigator, study coordinator or nurse). This evaluation was a general, aggregate assessment and was not linked to any specific participant. To assess Humalog Tempo Pen and Tempo smart button device usefulness HCPs were asked: "It improved my confidence in making appropriate dosing decisions".
  HCPs were categorized based on their responses on a 5-point Likert scale as below and are reported.
  1. Strongly Disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree
Time Frame: Following completion of participant's Last visit in the study (approximately 3 days after last visit on week 18)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 37
Participants
  Strongly Disagree | 1
  Disagree | 4
  Neutral | 15
  Agree | 13
  Strongly Agree | 4

24. Secondary Outcome: Health Care Provider (HCP) Questionnaires (Device Usefulness) - I Suspect That my Patients Miss Insulin Doses Regularly
Description: The Health Care Provider (HCP) questionnaires evaluated responses from HCPs related to Humalog Tempo Pen and Tempo smart button device focusing on satisfaction, preferences, and usefulness.
  Questionnaire was completed independently by HCPs (Including principal Investigator, study coordinator or nurse). This evaluation was a general, aggregate assessment and was not linked to any specific participant. To assess Humalog Tempo Pen and Tempo smart button device usefulness HCPs were asked: "I suspect that my patients miss insulin doses regularly".
  HCPs were categorized based on their responses on a 5-point Likert scale as below and are reported.
  1. Strongly Disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree
Time Frame: Following completion of participant's Last visit in the study (approximately 3 days after last visit on week 18)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 37
Participants
  Strongly Disagree | 4
  Disagree | 8
  Neutral | 19
  Agree | 5
  Strongly Agree | 1

25. Secondary Outcome: Health Care Provider (HCP) Questionnaires (Device Usefulness)- Allowed me to Objectively Discuss Missed Doses or Mistimed Doses With my Patients
Description: The Health Care Provider (HCP) questionnaires evaluated responses from HCPs related to Humalog Tempo Pen and Tempo smart button device focusing on satisfaction, preferences, and usefulness.
  Questionnaire was completed independently by HCP (Including principal Investigator, study coordinator or nurse. This evaluation was a general, aggregate assessment and was not linked to any specific participant. To assess Humalog Tempo Pen and Tempo smart button device usefulness HCPs were asked: "Allowed me to objectively discuss missed doses or mistimed doses with my patients".
  HCPs were categorized based on their responses on a 5-point Likert scale as below and are reported.
  1. Strongly Disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree
Time Frame: Following completion of participant's Last visit in the study (approximately 3 days after last visit on week 18)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Humalog Tempo Pen With CGM Monitoring
Number analyzed (Participants) | 37
Participants
  Strongly Disagree | 2
  Disagree | 3
  Neutral | 10
  Agree | 15
  Strongly Agree | 7

ADVERSE EVENTS:
Time Frame: Baseline Up to Week 18
Description: All enrolled participants. Based on the planned safety analysis, adverse events were collected per the overall treatment period, irrespective of study period (Period 1 or Period 2).
Arm/Group | Humalog Tempo Pen With CGM Monitoring
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 3/36
Other Adverse Events (participants affected / at risk) | 7/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Humalog Tempo Pen With CGM Monitoring (N=36)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Humalog Tempo Pen With CGM Monitoring (N=36)
Bronchitis (Infections and infestations) | 2 (2)
Covid-19 (Infections and infestations) | 3 (3)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT05893797/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/97/NCT05893797/SAP_001.pdf